CLINICAL TRIAL: NCT02964507
Title: A Phase I/II Dose Escalation and Expansion Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of GSK525762 in Combination With Fulvestrant in Subjects With Hormone Receptor-positive/HER2-negative (HR+/HER2-) Advanced or Metastatic Breast Cancer
Brief Title: Dose Escalation and Expansion Study of GSK525762 in Combination With Fulvestrant in Participants With Hormone Receptor-positive (HR+)/Human Epidermal Growth Factor Receptor 2 Negative (HER2-) Advanced or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study has been terminated due to meeting protocol defined futility.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201973; 2016-003074-40 (EudraCT Number)
Record Dates: First submitted 2016-11-12; First posted 2016-11-16 (Estimated); Results first posted 2022-01-27 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Neoplasms
Keywords: GSK525762; HR+/HER2- advanced or metastatic breast cancer; mTPI
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — molibresib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GSK525762 + Fulvestrant (Phase I) (Experimental)
  Interventions: Drug: GSK525762; Drug: Fulvestrant
- GSK525762 + Fulvestrant (Phase II) (Experimental)
  Interventions: Drug: GSK525762; Drug: Fulvestrant
- Placebo + Fulvestrant (Phase II) (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Fulvestrant

INTERVENTIONS:
Drug: GSK525762 — GSK525762 will be administered.
  Arms: GSK525762 + Fulvestrant (Phase I); GSK525762 + Fulvestrant (Phase II)
Drug: Placebo — Placebo will be administered.
  Arms: Placebo + Fulvestrant (Phase II)
Drug: Fulvestrant — Fulvestrant will be administered.

SUMMARY:
This is a combination Phase I and Phase II study, with an aim to evaluate the combination of GSK525762 and fulvestrant in women with HR+/HER2- advanced or metastatic breast cancer, who have disease that has progressed after prior treatment with at least one line of endocrine therapy. The objectives of the study are to first identify, in open-label single-arm Phase I, a recommended Phase II dose of GSK525762 that may be combined safely with fulvestrant. Phase I will follow a modified toxicity probability interval (mTPI) design, and a sentinel group will be evaluated first for dose-limiting toxicity and further expanded to collect additional safety data. This will be followed by a double-blind, randomized controlled Phase II, to identify the clinical activity of the two study treatments when given in combination. The composition of Phase II will be selected at the end of Phase I.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided.
* Females 18 years old and greater (at the time of written consent)
* Histologically or cytologically confirmed diagnosis of advanced or metastatic adenocarcinoma of the breast.
* Documentation of estrogen receptor (ER)-positive and/or progesterone receptor (PR)-positive tumor (>=1% positive stained tumor cell nuclei) based on local testing of the most recent tumor biopsy, using an assay consistent with local standards.
* Documentation of HER2-negative tumor based on local testing of the most recent tumor biopsy as per most recent American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines. At the time of writing, HER2-negative tumor is defined as immunohistochemistry (IHC) score of 0 or 1+, or negative by in situ hybridization defined as a HER2/chromosome enumeration probe 17 (CEP17) ratio <2 or for single probe assessment of an average HER2 copy number <4.
* Provision of mandatory screening fresh tumor biopsy sample during the screening period: a. Screening biopsy can be waived if a biopsy was collected within 3 months prior to first dose of study drug and was collected after the last anti-cancer treatment before coming into this study; b. Participants with inaccessible site of biopsy or who have a significant medical risk of obtaining the biopsy should be discussed with the Medical Monitor if they can qualify; c. Bone biopsies are not acceptable. Biopsies should be obtained from bone with metastatic soft-tissue component. Participants with bone only disease may be enrolled upon review by Medical Monitor.
* History of prior therapy that satisfies one of the following criteria: a. Aromatase inhibitor (AI) failures: Disease that relapsed during treatment or within 12 months of completion of adjuvant therapy with an AI, OR disease that progressed during treatment with an AI for advanced/metastatic disease. Prior ovarian suppression and/or tamoxifen are allowed as long as other criteria are met; b. Cyclin-dependent kinase 4/6 (CDK4/6) inhibitor plus AI failures: Disease that progressed on a CDK4/6 inhibitor plus AI, for advanced/metastatic disease with a minimum duration of treatment of 12 months (>=12 months) with CDK4/6 inhibitor plus AI. Participants with either measurable disease or bone only disease are allowed. Prior ovarian suppression and/or tamoxifen are allowed as long as other criteria are met.
* Documented progression on last line of systemic anti-cancer therapy with CDK4/6 inhibitor plus AI is required.
* Any menopausal status.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria is required except for participants with bone only disease.
* All prior treatment- related toxicities must be National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4 <=Grade 1 (except alopecia (permitted at any grade) and peripheral neuropathy (permitted at <=Grade 2) at the time of treatment allocation.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 to 1.
* Adequate organ function.
* Able to swallow and retain orally administered medication.
* A female participant is eligible to participate if she is of: i) Non-childbearing potential. ii) Child-bearing potential and agrees to use one of the contraception methods. iii) Negative serum pregnancy test <=7 days prior to first study drug dose. iv) Female participants who are lactating must discontinue nursing prior to the first dose of study treatment and must refrain from nursing throughout the treatment period and for at least 28 days following the last dose of study treatment.

Exclusion Criteria:

* Prior therapy with any Bromodomain and extra-terminal (BET) inhibitor, any selective estrogen receptor degrader (SERD) including fulvestrant, or inhibitors of the Phosphoinositide-3-kinase (PI3K)/ serine/threonine-specific protein kinase (AKT)/Mammalian Target of Rapamycin (mTOR) pathway.
* Prior therapy with more than one line of cytotoxic chemotherapy following diagnosis of advanced/metastatic disease.
* More than or equal to 3 lines of systemic anti-cancer therapy in the advanced or metastatic setting.
* Recent prior therapy, defined as: a. Any investigational or approved non-biologic anti-cancer drug within 14 days or five half-life (whichever is greater) prior to the first dose of GSK525762 and fulvestrant. b. Any nitrosoureas or mitomycin C within 42 days prior to the first dose of GSK525762 and fulvestrant c. Any anti-cancer biologic agents within 42 days prior to the first dose of GSK525762 and fulvestrant. d. Any radiotherapy within 14 days prior to the first dose of GSK525762 and fulvestrant. If the participant received radiotherapy <90 days prior to study treatment, the irradiated lesion cannot be the only lesion used for evaluating response.

  e. Any major surgery within 28 days prior to the first dose of GSK525762 and fulvestrant
* Concomitant active malignancy other than HR+/HER2- breast cancer
* Therapeutic-dose anticoagulation (e.g., warfarin, low-molecular weight heparin [LMWH], or novel oral anticoagulants) must be discontinued and coagulation parameters must be normalized prior to the first dose of GSK525762 and fulvestrant. Prophylactic anticoagulation, with low doses (per standard practice) of agents such as LMWH, direct thrombin inhibitors, or factor Xa inhibitors is permitted.
* Current use of a prohibited medication or planned use of any forbidden medications during treatment with GSK525762 and fulvestrant. This includes medications with significant risk of Torsades de pointes as well as those that are potent inducers or inhibitors of Cytochrome P3A4 (CYP3A4) enzymes.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, cardiac disease, or clinically significant bleeding episodes). Any serious and/or unstable pre-existing medical (aside from malignancy), psychiatric disorder, or other conditions that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator. a) Systolic blood pressure higher than 150 millimeters of mercury (mmHg) or diastolic blood pressure higher than 90 mmHg found on 2 separate occasions separated by 1 week, despite adequate therapy, will be defined as uncontrolled hypertension. b) Uncontrolled diabetes mellitus (despite therapeutic; compliance to intervention) as defined by a hemoglobin A1c (HbA1c) level more than 8% and/or occurrence of more than two episodes of ketoacidosis in the 12 months prior to the first dose of study drug.
* Participants with advanced/metastatic, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term including participants with massive uncontrolled effusions (pleural, pericardial, peritoneal), pulmonary lymphangitis, and over 50 percent (%) of liver involvement in metastases.
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression.
* Cardiac abnormalities as evidenced by any of the following: Baseline QT interval corrected by Fridericia's formula (QTcF) interval >=480 milliseconds (msec); Clinically significant conduction abnormalities or arrhythmias; Presence of cardiac pacemaker or defibrillator with a paced ventricular rhythm limiting electrocardiogram analysis; History or evidence of current >=Class II congestive heart failure as defined by New York Heart Association (NYHA); History of acute coronary syndromes (including unstable angina and myocardial infarction), coronary angioplasty, or stenting within the past 3 months. Participants with a history of stent placement requiring ongoing antithrombotic therapy (e.g., clopidogrel, prasugrel) will not be permitted to enroll; Clinically significant cardiomegaly, ventricular hypertrophy, or cardiomyopathy.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator assessment).
* Presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening.
* History of known human immunodeficiency virus (HIV) infection.
* Any serious known immediate or delayed hypersensitivity reaction(s) to GSK525762 or fulvestrant, or idiosyncrasy to drugs chemically related to the investigational drugs.
* Hemoptysis >1 teaspoon in 24 hours within the last 28 days.
* Concurrent use of non-steroidal anti-inflammatory drugs (NSAIDs) (except for cases where NSAIDs provide benefit over other analgesics and in these cases, consideration should be given to the prophylactic administration of a proton pump inhibitor) and high dose aspirin (allowed up to <=100 milligrams orally daily).
* Participants with history of known bleeding disorder(s) including clinically significant hemorrhage (e.g., gastrointestinal, neurologic), within the past 6 months.
* Any clinically significant gastrointestinal abnormalities that may alter absorption, such as malabsorption syndrome, chronic gastrointestinal disease, or major resection of the stomach and/or bowels that could preclude adequate absorption of the study medication.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 124 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2021-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- United States (15):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, White Plains, New York
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Seattle, Washington
- Australia (3):
  - GSK Investigational Site, Port Macquarie, New South Wales
  - GSK Investigational Site, Bedford Park, South Australia
  - GSK Investigational Site, Heidelberg, Victoria
- Canada (4):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- France (2):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Saint-Herblain
- South Korea (2):
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (3):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Lleida
- United Kingdom (5):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Nottingham, Nottinghamshire
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase I/II study of GSK525762 in combination with fulvestrant in participants with hormone receptor-positive/HER2-negative (HR+/HER2-)advanced/metastatic breast cancer. Out of 124 participants enrolled in the study, 1 participant was not treated.
Pre-assignment Details: As per study protocol, an interim analysis was conducted during phase 1,following assessment of data,phase 2 was not initiated. However,all existing participants receiving treatment in phase 1 who were considered to be deriving benefit were continued on the study (at investigators decision),until progression or death/withdrawal.As per the protocol the study was considered as completed when the last participant completed/discontinued study treatment and completed the end of treatment visit
Groups:
- Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure): Participants with aromatose inhibitor (AI) failure received GSK525762 60 milligrams (mg) tablet orally once daily and Fulvestrant (FUL) 500 mg was administered intramuscularly (IM) on days 1, 15, 29, and once monthly thereafter.
- Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M): Participants with Cyclin-Dependent Kinase (CDK4/6)/AI failure within 12 months received GSK525762 60 mg tablet orally once daily and FUL 500 mg was administered IM on days 1, 15, 29, and once monthly thereafter.
- Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M): Participants with CDK4/6/AI failure >=12 months received GSK525762 60 mg tablet orally once daily and FUL 500 mg was administered IM on days 1, 15, 29, and once monthly thereafter.
- Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease: Participants with CDK4/6/AI failure >=12 months with bone only disease received GSK525762 60 mg tablet orally once daily and FUL 500 mg was administered IM on days 1, 15, 29, and once monthly thereafter.
- Phase I-GSK525762 80mg + FUL 500 mg (AI Failure): Participants with AI failure received GSK525762 80 mg tablet orally once daily and FUL 500 mg was administered IM on days 1, 15, 29, and once monthly thereafter.
- Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure): Participants with CDK4/6/AI failure received GSK525762 80 mg tablet orally once daily and FUL 500 mg was administered IM on days 1, 15, 29, and once monthly thereafter.
- Phase II-GSK525762+FUL: Participants were planned to receive GSK525762+ FUL. The dose was to be decided based on the totality of the data at the end of Phase I.
- Phase II-Placebo+FUL: Participants were planned to receive Placebo+FUL. The dose was to be decided based on the totality of the data at the end of Phase I.
Period: Overall Study
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure) | Phase II-GSK525762+FUL | Phase II-Placebo+FUL
Started | 33 | 12 | 42 | 7 | 18 | 11 | 0 | 0
Completed | 7 | 1 | 17 | 1 | 2 | 3 | 0 | 0
Not Completed | 26 | 11 | 25 | 6 | 16 | 8 | 0 | 0
Not completed — Protocol specified Withdrawal criteria met | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Study terminated by Sponsor | 9 | 1 | 9 | 3 | 3 | 2 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 11 | 9 | 12 | 2 | 10 | 5 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 3 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The interim analysis failed to demonstrate clinically meaningful activity, hence Phase II was not initiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure) | Phase II-GSK525762+FUL | Phase II-Placebo+FUL | Total
Number analyzed (Participants) | 33 | 12 | 42 | 7 | 18 | 11 | 0 | 0 | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.6 (9.40) | 53.3 (8.48) | 55.7 (9.82) | 58.7 (7.97) | 54.4 (8.45) | 51.5 (12.04) |  |  | 56.4 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 12 | 42 | 7 | 18 | 11 | 0 | 0 | 123
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Central south Asian Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  East Asian Heritage | 7 | 2 | 8 | 1 | 6 | 2 | 0 | 0 | 26
  Japanese Heritage | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  South East Asian Heritage | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Black or African American | 2 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 8
  Arabic/North African Heritage | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3
  White/Caucasian/European Heritage | 19 | 8 | 28 | 5 | 11 | 7 | 0 | 0 | 78
  Multiple | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Missing | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, any other situation such as important medical events according to medical or scientific judgement or is associated with liver injury and impaired liver function. Any other adverse event apart from SAE is considered as non-SAE.
Time Frame: Up to 3 year and 8 months
Population: All Treated Population consisted of participants who received at least one dose of study treatment (GSK525762 or fulvestrant).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 33 | 12 | 42 | 7 | 18 | 11
Participants
  Non-serious AEs | 33 | 12 | 42 | 7 | 18 | 11
  SAEs | 5 | 1 | 10 | 3 | 6 | 2

2. Primary Outcome: Phase I: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: An event was considered DLT if it occurred within first 28 days of treatment and met one of following DLT criteria: Grade3 or greater neutropenia for >=5 days, febrile neutropenia, Grade4 anemia of any duration, Grade4 thrombocytopenia of any duration or Grade3 thrombocytopenia with bleeding, alanine aminotransferase (ALT) >3 times (x) upper limit of normal (ULN)+bilirubin >=2x ULN (>35 % direct) or ALT between 3-5xULN with bilirubin <2xULN but with hepatitis symptoms or rash, Grade3 nausea,vomiting or diarrhea that did not improve within 72hour despite appropriate supportive treatment(s), Grade4 nausea,vomiting,or diarrhea, Grade3 hypertension (uncontrolled despite addition of upto 2 antihypertensive medications), Grade4 hypertension, other Grade3 or greater clinically significant non-hematologic toxicity (including QT duration corrected for heart rate by Fridericia's formula (QTcF), ejection fraction <lower limit of normal (LLN) with an absolute decrease of >10% from Baseline.
Time Frame: Up to 28 days
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 33 | 12 | 42 | 7 | 18 | 11
Participants | 2 | 0 | 1 | 1 | 0 | 2

3. Primary Outcome: Phase I: Number of Participants With Dose Reductions and Dose Interruption/Delays
Description: Number of participants with dose reductions and dose interruption or delay due to any reason is presented.
Time Frame: Up to 3 year and 8 months
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 33 | 12 | 42 | 7 | 18 | 11
Participants
  Dose reduction | 9 | 3 | 14 | 3 | 7 | 8
  Dose interruption/delay | 23 | 9 | 23 | 4 | 15 | 9

4. Primary Outcome: Phase I: Objective Response Rate-Investigator Assessment
Description: Objective Response Rate is defined as the percentage of participants who demonstrate a Best Response of confirmed complete response (CR) or partial response (PR), as assessed by the investigator per response evaluation criteria in solid tumors (RECIST) version (v) 1.1 criteria.
Time Frame: Up to 3 year and 8 months
Population: Modified All Treated Population consisted of all participants who received at least one dose of GSK525762 and fulvestrant.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 33 | 12 | 42 | 7 | 18 | 11
Percentage of participants | 21 [9.0 to 38.9] | 0 [0.0 to 26.5] | 12 [4.0 to 25.6] | 0 [0.0 to 41.0] | 17 [3.6 to 41.4] | 9 [0.2 to 41.3]

5. Primary Outcome: Phase I: Plasma Concentration of GSK525762
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK525762.
Time Frame: Day 1: Pre-dose, 0.5, 1, 3 hours on Weeks 1 and 3; Day 1: Pre-dose, 0.5-1, 4-8 hours on Week 5; Day 1: Pre-dose, 0.5-1 hour on Weeks 9, 17, 25
Population: PK Population comprised of participants from the All Treated Population for whom a PK sample was obtained and analyzed. Only those participants with data available at the indicated time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 31 | 12 | 41 | 7 | 18 | 11
Nanograms per milliliter
  Week 1 Day 1, Pre-dose, n=30,11,41,7,17,11: number analyzed (Participants) | 30 | 11 | 41 | 7 | 17 | 11
  Week 1 Day 1, Pre-dose, n=30,11,41,7,17,11 | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose
  Week 1 Day 1, 0.5 hour, n=31,11,40,7,17,10: number analyzed (Participants) | 31 | 11 | 40 | 7 | 17 | 10
  Week 1 Day 1, 0.5 hour, n=31,11,40,7,17,10 | 895.466 (520.7900) | 814.364 (465.7197) | 824.081 (605.1745) | 646.251 (537.3585) | 969.265 (659.5862) | 1155.300 (329.8983)
  Week 1 Day 1, 1 hour, n=31,10,40,7,18,10: number analyzed (Participants) | 31 | 10 | 40 | 7 | 18 | 10
  Week 1 Day 1, 1 hour, n=31,10,40,7,18,10 | 855.734 (374.3789) | 828.800 (216.0544) | 947.343 (443.7234) | 634.300 (331.3116) | 1061.722 (397.9207) | 1069.400 (269.4864)
  Week 1 Day 1, 3 hours, n=31,10,39,6,17,10: number analyzed (Participants) | 31 | 10 | 39 | 6 | 17 | 10
  Week 1 Day 1, 3 hours, n=31,10,39,6,17,10 | 637.097 (220.5013) | 526.400 (106.3591) | 717.769 (293.5412) | 732.833 (394.3660) | 831.176 (293.0363) | 782.600 (191.9283)
  Week 3 Day 1, Pre-dose, n=29,12,31,5,16,8: number analyzed (Participants) | 29 | 12 | 31 | 5 | 16 | 8
  Week 3 Day 1, Pre-dose, n=29,12,31,5,16,8 | 7.046 (8.2049) | 15.797 (20.7736) | 8.598 (13.2639) | 150.410 (295.0514) | 11.371 (17.8450) | 6.799 (5.7108)
  Week 3 Day 1, 0.5 hour, n=28,11,29,4,13,7: number analyzed (Participants) | 28 | 11 | 29 | 4 | 13 | 7
  Week 3 Day 1, 0.5 hour, n=28,11,29,4,13,7 | 766.179 (330.0370) | 680.936 (435.2668) | 504.516 (342.6658) | 730.250 (410.6356) | 808.846 (548.7639) | 917.714 (498.7183)
  Week 3 Day 1, 1 hour, n=28,11,30,5,13,7: number analyzed (Participants) | 28 | 11 | 30 | 5 | 13 | 7
  Week 3 Day 1, 1 hour, n=28,11,30,5,13,7 | 737.536 (310.4540) | 576.427 (298.5082) | 581.073 (273.6803) | 596.800 (134.6540) | 875.077 (343.5570) | 895.286 (358.3172)
  Week 3 Day 1, 3 hours, n=28,10,29,5,13,7: number analyzed (Participants) | 28 | 10 | 29 | 5 | 13 | 7
  Week 3 Day 1, 3 hours, n=28,10,29,5,13,7 | 423.500 (190.6163) | 447.700 (179.1889) | 369.179 (171.4981) | 422.800 (120.6512) | 471.154 (160.2908) | 523.714 (207.9308)
  Week 5 Day 1, Pre-dose, n=26,9,34,5,14,10: number analyzed (Participants) | 26 | 9 | 34 | 5 | 14 | 10
  Week 5 Day 1, Pre-dose, n=26,9,34,5,14,10 | 5.804 (7.7777) | 15.251 (18.1145) | 66.527 (198.8847) | 15.814 (21.5282) | 14.603 (17.0653) | 77.465 (217.4469)
  Week 5 Day 1, 0.5-1 hour, n=24,7,26,3,11,7: number analyzed (Participants) | 24 | 7 | 26 | 3 | 11 | 7
  Week 5 Day 1, 0.5-1 hour, n=24,7,26,3,11,7 | 640.700 (380.5152) | 463.854 (476.0195) | 555.237 (336.1938) | 705.667 (208.2218) | 685.773 (446.6621) | 457.229 (301.9096)
  Week 5 Day 1, 4-8 hours, n=6,1,9,1,5,0: number analyzed (Participants) | 6 | 1 | 9 | 1 | 5 | 0
  Week 5 Day 1, 4-8 hours, n=6,1,9,1,5,0 | 306.900 (153.8008) | 145.000 (NA) — Standard deviation could not be calculated due to single participant | 303.000 (177.1489) | 431.000 (NA) — Standard deviation could not be calculated due to single participant | 352.400 (98.5890) |
  Week 9 Day 1, Pre-dose, n=17,2,23,2,10,4: number analyzed (Participants) | 17 | 2 | 23 | 2 | 10 | 4
  Week 9 Day 1, Pre-dose, n=17,2,23,2,10,4 | 7.257 (11.2876) | 5.055 (0.7142) | 9.000 (13.3106) | 3.265 (NA) — Standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than [>] 30 percent [%] of values were imputed). | 16.469 (23.7102) | 6.640 (7.0298)
  Week 9 Day 1, 0.5-1 hour, n=13,1,17,2,6,3: number analyzed (Participants) | 13 | 1 | 17 | 2 | 6 | 3
  Week 9 Day 1, 0.5-1 hour, n=13,1,17,2,6,3 | 607.408 (528.6891) | 69.400 (NA) — Standard deviation could not be calculated due to single participant | 445.291 (388.9562) | 817.000 (287.0854) | 621.867 (440.4829) | 309.627 (375.4223)
  Week 17 Day 1, Pre-dose, n=11,2,8,2,6,3: number analyzed (Participants) | 11 | 2 | 8 | 2 | 6 | 3
  Week 17 Day 1, Pre-dose, n=11,2,8,2,6,3 | 9.401 (13.0880) | 1.365 (NA) — Standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than [>] 30 percent [%] of values were imputed). | 3.591 (NA) — Standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than [>] 30 percent [%] of values were imputed). | 16.850 (2.0506) | 7.217 (10.1456) | 7.270 (NA) — Standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than [>] 30 percent [%] of values were imputed).
  Week 17 Day 1, 0.5-1 hour, n=9,2,9,2,4,1: number analyzed (Participants) | 9 | 2 | 9 | 2 | 4 | 1
  Week 17 Day 1, 0.5-1 hour, n=9,2,9,2,4,1 | 372.778 (214.7812) | 32.100 (30.2642) | 521.241 (404.3103) | 270.000 (354.9676) | 640.000 (273.7846) | 214.000 (NA) — Standard deviation could not be calculated due to single participant
  Week 25 Day 1, Pre-dose, n=9,1,5,2,4,1: number analyzed (Participants) | 9 | 1 | 5 | 2 | 4 | 1
  Week 25 Day 1, Pre-dose, n=9,1,5,2,4,1 | 34.847 (92.3723) | NA (NA) — No concentration values were detected for pre-dose | 10.198 (10.4909) | 10.740 (9.1358) | 1.560 (NA) — Standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than [>] 30 percent [%] of values were imputed). | NA (NA) — No concentration values were detected for pre-dose
  Week 25 Day 1, 0.5-1 hour, n=5,0,6,2,2,1: number analyzed (Participants) | 5 | 0 | 6 | 2 | 2 | 1
  Week 25 Day 1, 0.5-1 hour, n=5,0,6,2,2,1 | 418.000 (173.5439) |  | 380.483 (338.1430) | 251.350 (225.7792) | 314.000 (90.5097) | 186.000 (NA) — Standard deviation could not be calculated due to single participant

6. Primary Outcome: Phase II: Progression Free Survival (PFS)
Description: PFS is defined as the time (in months) from the date of first dose until the date of first documented progressive disease (PD), as assessed by the investigator per RECIST v1.1 criteria, or date of death due to any cause, whichever occurs first. PD is defined as at least a 20% increase in the sum of the diameters of target lesions taking as a reference the smallest sum of diameters for this study.
Time Frame: Up to 3 year and 8 months
Population: Modified All Treated Population. Phase II of study was not initiated hence data was not collected and analyzed.
Arm/Group | Phase II-GSK525762+FUL | Phase II-Placebo+FUL
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Phase I: Number of Participants Who Withdrew Due to Toxicity and Changes in Safety Assessment
Description: Number of participants who withdrew due to toxicity and changes in safety assessment including laboratory parameters and vital signs have been presented.
Time Frame: Up to 4 year and 4 months
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 33 | 12 | 42 | 7 | 18 | 11
Participants | 6 | 0 | 6 | 2 | 1 | 2

8. Secondary Outcome: Phase I: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants in the population with a confirmed complete response (CR), confirmed partial response (PR), or stable disease (SD) lasting >=6 months, as assessed by the investigator per RECIST v1.1 criteria.
Time Frame: Up to 3 year and 8 months
Population: Modified All Treated Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 33 | 12 | 42 | 7 | 18 | 11
Percentage of participants | 36 [20.4 to 54.9] | 0 [0.0 to 26.5] | 17 [7.0 to 31.4] | 14 [0.4 to 57.9] | 28 [9.7 to 53.5] | 9 [0.2 to 41.3]

9. Secondary Outcome: Phase I: Duration of Response (DoR)
Description: DoR is defined as the time (in months) from date of first documented evidence of confirmed CR or PR to the date of first documented PD, as assessed by the investigator per RECIST v1.1 criteria, or to the date of death due to any cause among participants with a Best overall response (BOR) of confirmed CR or PR.
Time Frame: Up to 3 year and 8 months
Population: Modified All Treated Population. Only those participants with a BOR of confirmed CR or PR based on RECIST v1.1 were analyzed hence N=0 for Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) and Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease arms.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 7 | 0 | 5 | 0 | 3 | 1
Months | 13.1 [6.5 to 26.3] |  | 5.8 [5.7 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. |  | 14.0 [5.4 to 16.4] | 4.3 [NA to NA] — Inter-quartile range is not applicable due to single participant, and the median value presented here is the actual DOR for this single participant

10. Secondary Outcome: Phase I: Progression-free Survival (PFS)
Description: PFS is defined as the time (in months) from the date of first dose until the date of first documented PD, as assessed by the investigator per RECIST v1.1 criteria, or date of death due to any cause, whichever occurs first. PD is defined as at least a 20% increase in the sum of the diameters of target lesions taking as a reference the smallest sum of diameters for this study.
Time Frame: Up to 3 year and 8 months
Population: Modified All Treated Population.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 33 | 12 | 42 | 7 | 18 | 11
Months | 5.6 [3.5 to 14.1] | 1.7 [1.6 to 2.1] | 2.1 [1.7 to 7.1] | 7.2 [3.7 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | 4.0 [1.8 to 9.4] | 1.8 [1.7 to 3.6]

11. Secondary Outcome: Phase I: Plasma Concentration of GSK3529246
Description: Blood samples were collected at indicated time points for PK analysis of GSK3529246. GSK3529246 is an active metabolite of GSK525762.
Time Frame: Day 1: Pre-dose, 0.5, 1, 3 hours on Weeks 1 and 3; Day 1: Pre-dose, 0.5-1, 4-8 hours on Week 5, Day 1: pre-dose, 0.5-1 hour on Weeks 9, 17, 25
Population: PK Population. Only those participants with data available at the indicated time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 31 | 12 | 41 | 7 | 18 | 11
Nanograms per milliliter
  Week 1 Day 1, Pre-dose, n=30,11,41,7,17,11: number analyzed (Participants) | 30 | 11 | 41 | 7 | 17 | 11
  Week 1 Day 1, Pre-dose, n=30,11,41,7,17,11 | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose
  Week 1 Day 1, 0.5 hour, n=31,11,39, 7,17,10: number analyzed (Participants) | 31 | 11 | 39 | 7 | 17 | 10
  Week 1 Day 1, 0.5 hour, n=31,11,39, 7,17,10 | 174.474 (143.3693) | 126.818 (84.5894) | 135.012 (128.9738) | 115.419 (108.8723) | 202.224 (225.2895) | 186.970 (108.3133)
  Week 1 Day 1, 1 hour, n=31,11,41,7,18,10: number analyzed (Participants) | 31 | 11 | 41 | 7 | 18 | 10
  Week 1 Day 1, 1 hour, n=31,11,41,7,18,10 | 249.793 (128.5670) | 205.364 (70.6856) | 228.597 (118.1550) | 175.197 (154.0632) | 327.072 (186.8822) | 299.100 (92.9043)
  Week 1 Day 1, 3 hours, n=31,11,39,6,17,10: number analyzed (Participants) | 31 | 11 | 39 | 6 | 17 | 10
  Week 1 Day 1, 3 hours, n=31,11,39,6,17,10 | 276.516 (67.1798) | 216.364 (50.0685) | 262.044 (91.2467) | 243.517 (136.5840) | 365.059 (130.8231) | 300.000 (95.1595)
  Week 3 Day 1, Pre-dose, n=29,12,31,5,16,8: number analyzed (Participants) | 29 | 12 | 31 | 5 | 16 | 8
  Week 3 Day 1, Pre-dose, n=29,12,31,5,16,8 | 37.972 (31.9814) | 58.708 (64.1009) | 42.213 (30.7403) | 121.820 (190.5127) | 48.013 (39.6626) | 49.230 (40.3798)
  Week 3 Day 1, 0.5 hour, n=28,11,30,4,13,7: number analyzed (Participants) | 28 | 11 | 30 | 4 | 13 | 7
  Week 3 Day 1, 0.5 hour, n=28,11,30,4,13,7 | 290.482 (155.8106) | 243.736 (130.5650) | 195.037 (147.9176) | 192.275 (149.9568) | 256.669 (173.4439) | 288.671 (166.5404)
  Week 3 Day 1, 1 hour, n=28,11,30,5,13,7: number analyzed (Participants) | 28 | 11 | 30 | 5 | 13 | 7
  Week 3 Day 1, 1 hour, n=28,11,30,5,13,7 | 414.143 (118.8203) | 294.573 (102.1516) | 323.767 (169.5878) | 271.200 (145.3227) | 511.692 (196.3468) | 441.571 (140.2353)
  Week 3 Day 1, 3 hours, n=28,10,29,5,13,7: number analyzed (Participants) | 28 | 10 | 29 | 5 | 13 | 7
  Week 3 Day 1, 3 hours, n=28,10,29,5,13,7 | 369.821 (85.0124) | 341.500 (95.5118) | 321.404 (131.8554) | 252.000 (96.1587) | 438.692 (91.5946) | 403.571 (96.7348)
  Week 5 Day 1, Pre-dose, n=26,9,34,5,14,10: number analyzed (Participants) | 26 | 9 | 34 | 5 | 14 | 10
  Week 5 Day 1, Pre-dose, n=26,9,34,5,14,10 | 37.480 (32.2441) | 41.600 (24.1873) | 56.659 (70.2933) | 36.620 (26.8511) | 52.243 (44.0710) | 54.231 (57.2752)
  Week 5 Day 1, 0.5-1 hour, n=24,7,26,3,11,7: number analyzed (Participants) | 24 | 7 | 26 | 3 | 11 | 7
  Week 5 Day 1, 0.5-1 hour, n=24,7,26,3,11,7 | 270.979 (153.7445) | 237.614 (211.1272) | 211.846 (171.4081) | 170.800 (66.2851) | 295.518 (235.4897) | 203.486 (111.2642)
  Week 5 Day 1, 4-8 hours, n=6,1,9,1,5,0: number analyzed (Participants) | 6 | 1 | 9 | 1 | 5 | 0
  Week 5 Day 1, 4-8 hours, n=6,1,9,1,5,0 | 263.833 (52.9619) | 208.000 (NA) — Standard deviation could not be calculated due to single participant | 322.778 (166.2354) | 292.000 (NA) — Standard deviation could not be calculated due to single participant | 382.400 (98.2588) |
  Week 9 Day 1, Pre-dose, n=17,2,23,2,10,4: number analyzed (Participants) | 17 | 2 | 23 | 2 | 10 | 4
  Week 9 Day 1, Pre-dose, n=17,2,23,2,10,4 | 31.041 (28.3504) | 33.850 (19.4454) | 39.323 (40.8779) | 22.700 (NA) — Standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than [>] 30 percent [%] of values were imputed). | 58.890 (62.2330) | 69.625 (53.3875)
  Week 9 Day 1, 0.5-1 hour, n=13,1,17,2,6,3: number analyzed (Participants) | 13 | 1 | 17 | 2 | 6 | 3
  Week 9 Day 1, 0.5-1 hour, n=13,1,17,2,6,3 | 244.162 (189.0153) | 36.000 (NA) — Standard deviation could not be calculated due to single participant | 178.914 (148.8777) | 228.000 (140.0071) | 283.667 (177.1211) | 161.367 (113.1437)
  Week 17 Day 1, Pre-dose, n=11,2,8,2,6,3: number analyzed (Participants) | 11 | 2 | 8 | 2 | 6 | 3
  Week 17 Day 1, Pre-dose, n=11,2,8,2,6,3 | 41.445 (35.8541) | 21.450 (5.4447) | 21.214 (27.8382) | 72.450 (55.9321) | 44.483 (48.7589) | 84.600 (74.6129)
  Week 17 Day 1, 0.5-1 hour, n=9,2,9,2,4,1: number analyzed (Participants) | 9 | 2 | 9 | 2 | 4 | 1
  Week 17 Day 1, 0.5-1 hour, n=9,2,9,2,4,1 | 189.422 (146.0021) | 71.800 (66.7509) | 183.671 (149.1568) | 129.050 (135.6938) | 322.500 (237.0787) | 301.000 (NA) — Standard deviation could not be calculated due to single participant
  Week 25 Day 1, Pre-dose, n=9,1,5,2,4,1: number analyzed (Participants) | 9 | 1 | 5 | 2 | 4 | 1
  Week 25 Day 1, Pre-dose, n=9,1,5,2,4,1 | 65.756 (125.0011) | 30.100 (NA) — Standard deviation could not be calculated due to single participant | 49.700 (26.2679) | 64.500 (60.1041) | 20.508 (29.5669) | NA (NA) — No concentration values were detected for pre-dose
  Week 25 Day 1, 0.5-1 hour, n=5,0,6,2,2,1: number analyzed (Participants) | 5 | 0 | 6 | 2 | 2 | 1
  Week 25 Day 1, 0.5-1 hour, n=5,0,6,2,2,1 | 203.160 (192.2849) |  | 220.367 (195.6110) | 204.950 (164.1195) | 121.300 (90.0854) | 76.300 (NA) — Standard deviation could not be calculated due to single participant

12. Secondary Outcome: Phase I: Plasma Concentration of Fulvestrant
Description: Blood samples were collected at indicated time points for PK analysis of Fulvestrant.
Time Frame: Day 1: Pre-dose on Weeks 1, 3, 5, 9, 17, 25
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 30 | 11 | 40 | 7 | 17 | 11
Nanograms per milliliter
  Week 1 Day 1, Pre-dose, n=30,11,40,6,17,11: number analyzed (Participants) | 30 | 11 | 40 | 6 | 17 | 11
  Week 1 Day 1, Pre-dose, n=30,11,40,6,17,11 | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose | NA (NA) — No concentration values were detected for pre-dose
  Week 3 Day 1, Pre-dose, n=30,11,32,7,16,10: number analyzed (Participants) | 30 | 11 | 32 | 7 | 16 | 10
  Week 3 Day 1, Pre-dose, n=30,11,32,7,16,10 | 13.32481 (6.603131) | 9.42742 (3.584881) | 12.44415 (5.669148) | 11.34839 (2.085675) | 12.41568 (4.873113) | 10.25047 (3.121508)
  Week 5 Day 1, Pre-dose, n=25,9,31,5,16,10: number analyzed (Participants) | 25 | 9 | 31 | 5 | 16 | 10
  Week 5 Day 1, Pre-dose, n=25,9,31,5,16,10 | 19.82642 (6.917439) | 14.72467 (3.338039) | 16.51574 (5.957079) | 15.35394 (5.395372) | 16.87293 (8.018589) | 13.83940 (4.449118)
  Week 9 Day 1, Pre-dose, n=19,3,19,1,10,5: number analyzed (Participants) | 19 | 3 | 19 | 1 | 10 | 5
  Week 9 Day 1, Pre-dose, n=19,3,19,1,10,5 | 16.33764 (5.719390) | 13.05750 (4.266495) | 13.98242 (4.138764) | 20.43840 (NA) — Standard deviation could not be calculated due to single participant | 11.10370 (2.864192) | 11.84244 (4.615995)
  Week 17 Day 1, Pre-dose, n=15,2,6,1,6,3: number analyzed (Participants) | 15 | 2 | 6 | 1 | 6 | 3
  Week 17 Day 1, Pre-dose, n=15,2,6,1,6,3 | 16.70103 (5.826390) | 20.63475 (7.753497) | 13.62853 (1.536930) | 12.59940 (NA) — Standard deviation could not be calculated due to single participant | 12.81337 (3.550671) | 16.33830 (4.410823)
  Week 25 Day 1, Pre-dose, n=10,1,4,1,4,1: number analyzed (Participants) | 10 | 1 | 4 | 1 | 4 | 1
  Week 25 Day 1, Pre-dose, n=10,1,4,1,4,1 | 18.07473 (5.933472) | 14.21220 (NA) — Standard deviation could not be calculated due to single participant | 18.60548 (5.300211) | 19.05100 (NA) — Standard deviation could not be calculated due to single participant | 16.05110 (2.384935) | 12.24970 (NA) — Standard deviation could not be calculated due to single participant

13. Secondary Outcome: Phase II: Overall Survival (OS)
Description: OS is defined as the interval of time (in months) between the date of first dose and the date of death due to any cause.
Time Frame: Up to 3 year and 8 months
Population: Modified All Treated Population. Phase II of study was not initiated hence data was not collected and analyzed.
Groups:
- Phase II-GSK525762 +FUL: Participants were planned to receive GSK525762+ FUL. The dose was to be decided based on the totality of the data at the end of Phase I.
Arm/Group | Phase II-GSK525762 +FUL | Phase II-Placebo+FUL
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Phase II: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants in the population who demonstrate a BOR of confirmed CR or PR, as assessed by the investigator per RECIST v1.1 criteria.
Time Frame: Up to 3 year and 8 months
Population: Modified All Treated Population. Phase II of study was not initiated hence data was not collected and analyzed.
Arm/Group | Phase II-GSK525762 +FUL | Phase II-Placebo+FUL
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Phase II: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants in the population with a confirmed CR, confirmed PR, or SD lasting >=6 months, as assessed by the investigator per RECIST v1.1 criteria.
Time Frame: Up to 3 year and 8 months
Population: Modified All Treated Population. Phase II of study was not initiated hence data was not collected and analyzed.
Arm/Group | Phase II-GSK525762 +FUL | Phase II-Placebo+FUL
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Phase II: Plasma Concentration of GSK525762 and GSK3529246
Description: Blood samples were planned to be collected for PK analysis of GSK525762 and GSK3529246. GSK3529246 is metabolite of GSK525762.
Time Frame: as for outcome 11
Population: PK Population. Phase II of study was not initiated hence data was not collected and analyzed.
Arm/Group | Phase II-GSK525762 +FUL | Phase II-Placebo+FUL
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Phase II: Plasma Concentration of Fulvestrant
Description: Blood samples were planned to be collected for PK analysis of fulvestrant.
Time Frame: Day 1: Pre-dose on Weeks 1, 3, 5, 9, 17, 25
Population: PK Population. Phase II of study was not initiated hence data was not collected and analyzed.
Arm/Group | Phase II-GSK525762+FUL | Phase II-Placebo+FUL
Number analyzed (Participants) | 0 | 0

18. Other Pre Specified Outcome: Phase I: Number of Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs) Until End of the Study
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, any other situation such as important medical events according to medical or scientific judgement or is associated with liver injury and impaired liver function. Any other adverse event apart from SAE is considered as non-SAE. Number of participants with non-serious AEs and SAEs collected from start of the treatment until end of the study were reported.
Time Frame: Up to 4 year and 4 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 33 | 12 | 42 | 7 | 18 | 11
Participants
  Non-serious AEs | 33 | 12 | 42 | 7 | 18 | 11
  SAEs | 5 | 1 | 10 | 3 | 6 | 2

19. Other Pre Specified Outcome: Phase I: Number of Participants With Dose Reductions and Dose Interruption/Delays Until End of the Study
Description: Number of participants with dose reductions and dose interruption or delay due to any reason is presented. Number of participants with dose reductions and dose interruption or delay due to any reason from start of the treatment until end of the study were reported.
Time Frame: Up to 4 year and 4 months
Population: All Treated Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I-GSK525762 60 mg+FUL 500 mg (AI Failure) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+AI Failure <12M) | Phase I-GSK525762 60 mg+FUL 500 mg (CDK4/6+ AI Failure >= 12M) | Phase I-GSK525762 60+FUL500mg CDK4/6+AI Failure>=12M Bone Only Disease | Phase I-GSK525762 80mg + FUL 500 mg (AI Failure) | Phase I-GSK525762 80 mg + FUL 500 mg (CDK4/6+AI Failure)
Number analyzed (Participants) | 33 | 12 | 42 | 7 | 18 | 11
Participants
  Dose reduction | 9 | 3 | 14 | 3 | 7 | 8
  Dose interruption/delay | 23 | 9 | 23 | 4 | 15 | 9

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious and non-serious adverse events were collected up to 4 year and 4 months
Description: All Treated Population consisted of participants who received at least one dose of study treatment (GSK525762 or fulvestrant). The interim analysis failed to demonstrate clinically meaningful activity, hence Phase II was not initiated. Data is presented for Phase I as data was not collected for Phase II.
Groups:
- Phase I- GSK525762 60mg+FUL 500mg (AI Failure): Participants with aromatose inhibitor (AI) failure received GSK525762 60 milligrams (mg) tablet orally once daily and Fulvestrant (FUL) 500 mg was administered intramuscularly (IM) on days 1, 15, 29, and once monthly thereafter.
- Phase I-GSK525762 60mg+FUL 500mg (CDK4/6+AI Failure < 12M): Participants with Cyclin-Dependent Kinase (CDK4/6)/AI failure within 12 months received GSK525762 60 mg tablet orally once daily and FUL 500 mg was administered IM on days 1, 15, 29, and once monthly thereafter.
- Phase I-GSK525762 60mg+FUL 500mg (CDK4/6+AI Failure >=12M): Participants with CDK4/6/AI failure >=12 months received GSK525762 60 mg tablet orally once daily and FUL 500 mg was administered IM on days 1, 15, 29, and once monthly thereafter.
- Phase I-GSK525762 60mg+FUL 500mg (CDK4/6+AI Failure >=12M Bone Only Disease: Participants with CDK4/6/AI failure >=12 months with bone only disease received GSK525762 60 mg tablet orally once daily and FUL 500 mg was administered IM on days 1, 15, 29, and once monthly thereafter.
- Phase I-GSK525762 80mg+FUL 500mg (AI Failure): Participants with AI failure received GSK525762 80 mg tablet orally once daily and FUL 500 mg was administered IM on days 1, 15, 29, and once monthly thereafter.
- Phase I-GSK525762 80mg+FUL 500mg (CDK4/6+AI Failure): Participants with CDK4/6/AI failure received GSK525762 80 mg tablet orally once daily and FUL 500 mg was administered IM on days 1, 15, 29, and once monthly thereafter.
- Phase II-Placebo+FUL: Participants were planned to receive GSK525762+ FUL. The dose was to be decided based on the totality of the data at the end of Phase I.
Arm/Group | Phase I- GSK525762 60mg+FUL 500mg (AI Failure) | Phase I-GSK525762 60mg+FUL 500mg (CDK4/6+AI Failure < 12M) | Phase I-GSK525762 60mg+FUL 500mg (CDK4/6+AI Failure >=12M) | Phase I-GSK525762 60mg+FUL 500mg (CDK4/6+AI Failure >=12M Bone Only Disease | Phase I-GSK525762 80mg+FUL 500mg (AI Failure) | Phase I-GSK525762 80mg+FUL 500mg (CDK4/6+AI Failure) | Phase II-GSK525762 +FUL | Phase II-Placebo+FUL
All-Cause Mortality (participants affected / at risk) | 11/33 | 9/12 | 12/42 | 2/7 | 10/18 | 5/11 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 5/33 | 1/12 | 10/42 | 3/7 | 6/18 | 2/11 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 33/33 | 12/12 | 42/42 | 7/7 | 18/18 | 11/11 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I- GSK525762 60mg+FUL 500mg (AI Failure) (N=33) | Phase I-GSK525762 60mg+FUL 500mg (CDK4/6+AI Failure < 12M) (N=12) | Phase I-GSK525762 60mg+FUL 500mg (CDK4/6+AI Failure >=12M) (N=42) | Phase I-GSK525762 60mg+FUL 500mg (CDK4/6+AI Failure >=12M Bone Only Disease (N=7) | Phase I-GSK525762 80mg+FUL 500mg (AI Failure) (N=18) | Phase I-GSK525762 80mg+FUL 500mg (CDK4/6+AI Failure) (N=11) | Phase II-GSK525762 +FUL (N=0) | Phase II-Placebo+FUL (N=0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diaphragmatic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extramammary Paget's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I- GSK525762 60mg+FUL 500mg (AI Failure) (N=33) | Phase I-GSK525762 60mg+FUL 500mg (CDK4/6+AI Failure < 12M) (N=12) | Phase I-GSK525762 60mg+FUL 500mg (CDK4/6+AI Failure >=12M) (N=42) | Phase I-GSK525762 60mg+FUL 500mg (CDK4/6+AI Failure >=12M Bone Only Disease (N=7) | Phase I-GSK525762 80mg+FUL 500mg (AI Failure) (N=18) | Phase I-GSK525762 80mg+FUL 500mg (CDK4/6+AI Failure) (N=11) | Phase II-GSK525762 +FUL (N=0) | Phase II-Placebo+FUL (N=0)
Nausea (Gastrointestinal disorders) | 12 (17) | 7 (10) | 30 (38) | 5 (9) | 11 (21) | 9 (9) | 0 (0) | 0 (0)
Fatigue (General disorders) | 19 (24) | 4 (6) | 25 (38) | 1 (1) | 9 (12) | 7 (10) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 14 (16) | 2 (3) | 25 (30) | 4 (4) | 10 (14) | 7 (8) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 13 (19) | 4 (4) | 20 (28) | 6 (10) | 10 (24) | 4 (4) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 14 (18) | 2 (3) | 18 (19) | 3 (5) | 9 (15) | 6 (7) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (21) | 3 (3) | 16 (22) | 3 (5) | 6 (11) | 2 (5) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 6 (25) | 2 (3) | 12 (21) | 2 (5) | 6 (12) | 4 (6) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 15 (19) | 3 (4) | 6 (9) | 2 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (6) | 2 (2) | 8 (9) | 4 (7) | 10 (20) | 2 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (4) | 13 (17) | 2 (2) | 3 (4) | 4 (5) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 3 (4) | 10 (11) | 1 (1) | 7 (10) | 3 (5) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2) | 13 (15) | 1 (1) | 1 (2) | 3 (5) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 8 (10) | 4 (4) | 10 (11) | 1 (1) | 4 (7) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (7) | 2 (2) | 11 (15) | 3 (5) | 5 (10) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 3 (3) | 10 (12) | 3 (8) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (15) | 4 (4) | 8 (14) | 4 (8) | 3 (9) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (8) | 2 (3) | 8 (9) | 2 (2) | 7 (9) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 2 (2) | 4 (4) | 2 (2) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7) | 2 (2) | 6 (6) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (5) | 1 (1) | 6 (6) | 4 (4) | 3 (4) | 4 (4) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 8 (9) | 3 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 4 (5) | 0 (0) | 7 (8) | 2 (5) | 3 (6) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 4 (4) | 2 (2) | 3 (6) | 3 (3) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 8 (8) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 9 (9) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 2 (3) | 2 (3) | 4 (5) | 2 (3) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 8 (11) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 7 (8) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1) | 5 (6) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2) | 2 (3) | 1 (2) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 4 (6) | 1 (1) | 4 (5) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 1 (1) | 5 (7) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 4 (7) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (7) | 3 (4) | 1 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 5 (5) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 1 (1) | 3 (3) | 0 (0) | 1 (4) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 4 (4) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 4 (8) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 6 (10) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 2 (3) | 1 (2) | 3 (3) | 1 (1) | 1 (5) | 2 (6) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 5 (7) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 2 (4) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (7) | 0 (0) | 4 (6) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 3 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 (2) | 1 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (3) | 0 (0) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT02964507/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT02964507/SAP_001.pdf